CLINICAL TRIAL: NCT02817659
Title: A Pilot Study to Determine Tolerability to Glucagon Infusion in Obese Subjects
Brief Title: To Determine Tolerability to Glucagon Infusion in Obese Subjects
Acronym: GIO
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AdventHealth Translational Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TRIMDFH 778967
Record Dates: First submitted 2016-06-08; First posted 2016-06-29 (Estimated); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Obesity
Keywords: Glucagon
MeSH Terms: conditions — Obesity | interventions — Glucagon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Glucagon Infusion (Experimental): Glucagon infusion in escalating manner at 12.5, 25, 37.5 and 50 ng/kg/min (each step for 60 min). At 30 and 60 mins of each infusion rate, we will administer a previously established questionnaire to assess overall nausea intensity.
  Interventions: Drug: Glucagon

INTERVENTIONS:
Drug: Glucagon — Glucagon infusion

SUMMARY:
To further understand the tolerability of glucagon.

DETAILED DESCRIPTION:
To determine the tolerability of glucagon infusion administered in an escalating step-wise manner in healthy obese subjects

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-55 years, inclusive
2. BMI ≥27 to ≤40 kg/m2
3. Stable body weight for 3 months (self-reported loss/gain <5%)
4. Subject is judged to be non-diabetic and in good health on the basis of medical history, physical examination, electrocardiogram, and routine laboratory data
5. Subject understands the procedures and agrees to participate in the study program by giving written informed consent, and is willing to comply with the trial restrictions
6. Subject is willing to avoid alcohol consumption for 48 hours prior to the inpatient study visit
7. Subject is willing to avoid consumption of caffeine and caffeinated beverages for 24 hours prior to the inpatient study visit
8. Subject is willing to avoid strenuous physical activity for 72 hours prior to the inpatient study visit
9. Female subjects of child bearing potential must be willing to use acceptable birth control during study participation (oral contraceptives, intrauterine device, implanted or injectable contraceptives, abstinence).

Exclusion Criteria:

1. Treatment with any medication known to significantly impact body weight (e.g., weight loss medications, atypical antipsychotics) within 3 months prior to screening except for stable physiological hormone replacement therapy (i.e., thyroid hormone, estrogen)
2. History of bariatric surgery
3. Current liver, renal, pulmonary, cardiac, oncologic, metabolic, gastrointestinal or hematologic disease which the Investigator believes is clinically significant, including:

   1. Liver disease or liver injury as indicated by abnormal liver function tests (aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase , serum bilirubin) >3 × upper limit of normal (ULN), or history of hepatic cirrhosis
   2. History or presence of impaired renal function as indicated by an estimated glomerular filtration rate <60 ml/hr or urine albumin-to-creatinine ratio >35 mg/mmol
   3. Significant cardiovascular disease, including Class III or greater congestive heart failure (CHF), coronary artery disease, second degree or greater heart block, or clinically significant arrhythmias; baseline second degree or greater heart block or prolonged QT syndrome (QTc interval ≥ 470 msec); or any major cardiovascular event within the last 3 years (including myocardial infarction, transient ischemic attack [TIA], cerebrovascular accident [CVA], angina, and hospitalization due to CHF, transient ischemic attack (TIA), and CVA)
   4. Metabolic, other or endocrine disorders, including diagnosis of type 1 or type 2 diabetes mellitus [HbA1c ≥6.5%]), inadequately treated hyperthyroidism (thyroid stimulating hormone [TSH] below normal range) or hypothyroidism (TSH above upper limit of normal if symptomatic or TSH >10 U/mL), Cushing syndrome, Addison's disease, hypogonadism, or genetic disorders linked to obesity
   5. History of irritable bowel disease, recurrent nausea or vomiting
   6. Anemia (hemoglobin <12 g/dl in men, <11 g/dl in women)
4. Self-reported history of hepatitis B, hepatitis C, or HIV
5. History of recurrent sleep disturbances and/or prone to sleep disturbances based on lifestyle or employment (e.g., variable work schedule, overnight shift work, etc.)
6. Diagnosis of sleep apnea with or without use of (continuous positive airway pressure)
7. Major surgery within last 3 months
8. Blood donation within 4 weeks prior to the screening visit
9. Participation in another investigational trial within 4 weeks prior to the screening visit. The 4 week window will be derived from the date of the last trial medication and/or blood collection in a previous trial and/or adverse event (AE) related to trial drug to the screening visit of the current trial.
10. Illicit drug abuse or use of nicotine-containing products within 3 months prior to the screening visit
11. Poor intravenous access
12. Blood pressure less than 100/50 mm Hg or greater than or equal to 160/100 mm Hg at screening visit
13. Heart rate greater than or equal to 100 beats/min at screening visit
14. Fasting plasma glucose <60 mg/dL or ≥126 mg/dL at screening visit
15. Translational Research Institute (TRI) staff member or immediate relative of TRI staff member, directly involved with this study
16. History of any illness or condition that, in the opinion of the study investigator, might confound the results of the study or poses an additional risk to the subject by study participation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-01-13 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Measure glucagon tolerance in healthy obese subject prior to subject becoming significantly nauseous. | Visit 1, measured at 30 minutes
  Glucagon infused in escalating manner. Each dose administered for 60 minutes. Intensity of nausea measured by administering a questionnaire that measures overall nausea intensity.
Measure glucagon tolerance in healthy obese subject prior to subject becoming significantly nauseous. | Visit 1, measured at 60 minutes
  Glucagon infused in escalating manner. Each dose administered for 60 minutes. Intensity of nausea measured by administering a questionnaire that measures overall nausea intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Smith, MD, Principal Investigator — Prinicipal Investigator
Locations (1):
- Translational Research Institute for Metabolism and Diabetes, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Astrup A, Rossner S, Van Gaal L, Rissanen A, Niskanen L, Al Hakim M, Madsen J, Rasmussen MF, Lean ME; NN8022-1807 Study Group. Effects of liraglutide in the treatment of obesity: a randomised, double-blind, placebo-controlled study. Lancet. 2009 Nov 7;374(9701):1606-16. doi: 10.1016/S0140-6736(09)61375-1. Epub 2009 Oct 23. PMID 19853906
- [Background] Flint A, Raben A, Rehfeld JF, Holst JJ, Astrup A. The effect of glucagon-like peptide-1 on energy expenditure and substrate metabolism in humans. Int J Obes Relat Metab Disord. 2000 Mar;24(3):288-98. doi: 10.1038/sj.ijo.0801126. PMID 10757621
- [Background] Cryer PE. Minireview: Glucagon in the pathogenesis of hypoglycemia and hyperglycemia in diabetes. Endocrinology. 2012 Mar;153(3):1039-48. doi: 10.1210/en.2011-1499. Epub 2011 Dec 13. PMID 22166985
- [Background] SCHULMAN JL, CARLETON JL, WHITNEY G, WHITEHORN JC. Effect of glucagon on food intake and body weight in man. J Appl Physiol. 1957 Nov;11(3):419-21. doi: 10.1152/jappl.1957.11.3.419. No abstract available. PMID 13480952
- [Background] Nair KS. Hyperglucagonemia increases resting metabolic rate in man during insulin deficiency. J Clin Endocrinol Metab. 1987 May;64(5):896-901. doi: 10.1210/jcem-64-5-896. PMID 2881943
- [Background] Calles-Escandon J. Insulin dissociates hepatic glucose cycling and glucagon-induced thermogenesis in man. Metabolism. 1994 Aug;43(8):1000-5. doi: 10.1016/0026-0495(94)90180-5. PMID 8052138
- [Background] Salem V, Izzi-Engbeaya C, Coello C, Thomas DB, Chambers ES, Comninos AN, Buckley A, Win Z, Al-Nahhas A, Rabiner EA, Gunn RN, Budge H, Symonds ME, Bloom SR, Tan TM, Dhillo WS. Glucagon increases energy expenditure independently of brown adipose tissue activation in humans. Diabetes Obes Metab. 2016 Jan;18(1):72-81. doi: 10.1111/dom.12585. Epub 2015 Nov 20. PMID 26434748
- [Background] Melzack R, Rosberger Z, Hollingsworth ML, Thirlwell M. New approaches to measuring nausea. CMAJ. 1985 Oct 15;133(8):755-8, 761. PMID 4042058
- [Background] Tan TM, Field BC, McCullough KA, Troke RC, Chambers ES, Salem V, Gonzalez Maffe J, Baynes KC, De Silva A, Viardot A, Alsafi A, Frost GS, Ghatei MA, Bloom SR. Coadministration of glucagon-like peptide-1 during glucagon infusion in humans results in increased energy expenditure and amelioration of hyperglycemia. Diabetes. 2013 Apr;62(4):1131-8. doi: 10.2337/db12-0797. Epub 2012 Dec 17. PMID 23248172
- [Background] Miyoshi H, Shulman GI, Peters EJ, Wolfe MH, Elahi D, Wolfe RR. Hormonal control of substrate cycling in humans. J Clin Invest. 1988 May;81(5):1545-55. doi: 10.1172/JCI113487. PMID 3284915
- See also: Florida Hospital Translational Research Institute for Metabolism and Diabetes — http://www.tri-md.org